CLINICAL TRIAL: NCT04169711
Title: A Phase 1b Dose-Finding Study of ARO-HIF2 in Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: Study of ARO-HIF2 in Patients With Advanced Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AROHIF21001
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARO-HIF2 (Experimental)
  Interventions: Drug: ARO-HIF2

INTERVENTIONS:
Drug: ARO-HIF2 — Multiple doses of ARO-HIF2 by intravenous infusion

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ARO-HIF2 injection (also referred to as ARO-HIF2) and to determine the recommended Phase 2 dose in the treatment of patients with advanced clear cell renal cell carcinoma (ccRCC).

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* Histologically confirmed locally advanced or metastatic clear cell renal cell carcinoma that has progressed during or after at least two prior therapeutic regimens which must include vascular endothelial growth factor (VEGF)-targeted therapy and checkpoint inhibitor therapy or that has otherwise failed such therapies, is measurable disease per RECIST 1.1 criteria, is biopsy accessible
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Estimated life expectancy of longer than 3 months
* Adequate organ function at screening

Exclusion Criteria:

* History of untreated brain metastasis or leptomeningeal disease or spinal cord compression
* Failure to recover from reversible effects of prior anti-cancer therapy
* Has received systemic therapy or radiation therapy within 2 weeks prior to first dose
* History of solid organ or stem cell transplantation
* Current use of anti-VEGF or mammalian target of rapamycin (mTOR) agents, or chronic immunosuppressive therapy
* Any prior use of hypoxia inducible factor 2 (HIF2) inhibitors within 6 months prior to first dose
* Current use of immune checkpoint inhibitors
* Use of an investigational agent or device within 2 weeks prior to dosing, or current participation in an investigational study
* Known HIV, hepatitis B or hepatitis C
* History of other clinically meaningful disease
* Major surgery within 4 weeks of Screening
* Active malignancy requiring therapy other than ccRCC within 3 years of study entry

Note: Other eligibility criteria may apply per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) Possibly or Probably Related to Treatment | Up to 2 years from first dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-HIF2: Maximum Observed Plasma Concentration (Cmax) | Up to Week 2: predose and up to 48 hours postdose
PK of ARO-HIF2: Time to Maximum Plasma Concentration (Tmax) | Up to Week 2: predose and up to 48 hours postdose
PK of ARO-HIF2: Area Under the Plasma Concentration Versus Time Curve from Zero to 4 Hours (AUC0-4) | Up to Week 2: predose and up to 48 hours postdose
PK of ARO-HIF2: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Up to Week 2: predose and up to 48 hours postdose
PK of ARO-HIF2: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Measurable Concentration at a Time=t, Using a Specified Trapezoidal Rule (AUC0-t) | Up to Week 2: predose and up to 48 hours postdose
PK of ARO-HIF2: Area Under the Plasma Concentration Versus Time Curve from Zero to Infinity (AUCinf) | Up to Week 2: predose and up to 48 hours postdose
PK of ARO-HIF2: Terminal Elimination Half-Life (t1/2) | Up to Week 2: predose and up to 48 hours postdose
Systemic Clearance Derived From Intravenous Dose/Area Under the Plasma Concentration Versus Time Curve (CL) | Up to Week 2: predose and up to 48 hours postdose
Amount of Drug Excreted in the Urine Over One Dosing Interval Through 4 Hours Post- Dose (Ae, 0-4) | Up to Week 2: predose and up to 48 hours postdose
Renal Clearance Calculated by Ae, 0-4 h/AUC0-4h (CLR) | Up to Week 2: predose and up to 48 hours postdose
Fraction Excreted (or Equivalently the Percent of Dose Excreted) in the Urine, Calculated by 100 X (Ae, 0-4 h/Dose) | Up to Week 2: predose and up to 48 hours postdose
Overall Response Rate | Baseline until disease progression, up to 2 years
  Percentage of participants with a best overall response of complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 criteria.
Duration of Response | Baseline until disease progression, up to 2 years
Time to Response | Baseline until disease progression, up to 2 years
Progression Free Survival | up to 2 years
Overall Survival | up to 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site 1, Aurora, Colorado
  - Research Site 2, Las Vegas, Nevada
  - Research Site 4, Nashville, Tennessee
  - Research Site 5, Dallas, Texas
  - Research Site 6, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided